CLINICAL TRIAL: NCT03299088
Title: A Phase Ib Trial of Pembrolizumab (MK-3475) and Trametinib Focused on Advanced KRAS Mutant Non-small Cell Lung Cancer
Brief Title: Pembrolizumab and Trametinib in Treating Patients With Stage IV Non-Small Cell Lung Cancer and KRAS Gene Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonathan Riess (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Novartis (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jonathan Riess, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1099442; UCDCC#259 (Registry Identifier: UC Davis IRB); UCDCC#259 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2017-01633 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: KRAS Gene Mutation; Metastatic Non-Squamous Non-Small Cell Lung Carcinoma; Recurrent Non-Squamous Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (trametinib, pembrolizumab) (Experimental): Patients receive trametinib PO daily. Beginning on day 1 of course 2, patients also receive pembrolizumab IV over 30 minutes. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib
- Arm B (pembrolizumab, trametinib) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Beginning on day 1 of course 2, patients also receive trametinib PO daily. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Trametinib

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase Ib trial studies the side effects of pembrolizumab and trametinib in treating patients with non-small cell lung cancer and KRAS gene mutations that has spread to other places in the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and trametinib may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of pembrolizumab (MK-3475) when given in combination with trametinib in the proposed sequencing schemes in patients with advanced or metastatic non-small cell lung cancer with KRAS mutations.

SECONDARY OBJECTIVES:

To assess in a preliminary manner the clinical efficacy of these combinations with the proposed sequencing schemes including overall response rate and progression free survival.

TERTIARY OBJECTIVES:

To determine in an exploratory manner changes in PD-L1 expression as well as other immune correlates induced by mitogen-activated extracellular signal-regulated kinase (MEK) inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or metastatic/recurrent non-small cell lung cancer; for expansion cohorts, patient's tumor must also harbor a KRAS mutation detected in a CLIA certified laboratory
* Have histologically or cytologically confirmed non-small cell lung cancer
* Have stage IV, metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC) with progressive disease after platinum containing chemotherapy (EGFR mutant, ALK, or ROS-1 rearranged NSCLC must have progressed on prior approved tyrosine kinase inhibitor [TKI]'s)
* For phase I dose expansion cohorts the patient's tumor must harbor a KRAS mutation detected by a CLIA certified laboratory
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion; in the opinion of the investigator, the patient must have tumor accessible by CT or ultrasound guided core biopsy; subjects for whom newly-obtained samples cannot be provided may submit an archived specimen provided it was obtained after last systemic treatment, within 6 months of signing consent and that tissue is available for either 2 cell blocks or 20 uncut slides (core or excisional biopsy required, fine needle aspirate is not acceptable)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Absolute neutrophil count >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x upper limit of normal (ULN)
* Albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine =< 1.5 ULN
* Calculated creatinine clearance >= 50 mL/min
* Left ventricular ejection fraction (LVEF) >= lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition (MUGA)
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication; note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy; note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Clarification: subjects with atrial fibrillation controlled for > 30 days prior to dosing are eligible

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; inhaled or topical steroids are allowed
* Has a known history of active tuberculosis (TB [Bacillus Tuberculosis])
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 3 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 3 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; note: subjects with =< grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study; note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis; history of radiation pneumonitis is allowed provided that it is not active and no corticosteroids were required for pneumonitis management
* Evidence of interstitial lung disease
* Has an active infection requiring systemic therapy
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO)
* History of retinal vein occlusion (RVO)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent for dose expansion; (patients in dose escalation may have received an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent)
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Has known active Hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] is detected)
* LVEF < LLN on screening exam
* A QT interval corrected for heart rate using the Fridericia's formula (QTcF) >= 470 msec on screening exam
* History or evidence of current clinically significant uncontrolled arrhythmias
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrollment
* History or evidence of current >= class II congestive heart failure as defined by New York Heart Association (NYHA)
* Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy
* Patients with intra-cardiac defibrillators
* Has received a live vaccine within 30 days of planned start of study therapy; note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Riess, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Escalation Arm A Dose Level 1: Trametinib 1.5 mg PO D1-10, Pembrolizumab 200 mg administered D1 starting with C2, Q21 days
- Escalation Arm A Dose Level 2: Trametinib 2 mg PO D1-10, Pembrolizumab 200 mg administered D1 starting with C2, Q21 days
- Escalation Arm B Dose Level 1: Trametinib 1.5 mg PO D1-10 starting with C2, Pembrolizumab 200 mg administered D1, Q21 days
- Escalation Arm B Dose Level 2: Trametinib 2 mg PO D1-10 starting with C2, Pembrolizumab 200 mg administered D1, Q21 days
Period: Overall Study
Arm/Group | Escalation Arm A Dose Level 1 | Escalation Arm A Dose Level 2 | Escalation Arm B Dose Level 1 | Escalation Arm B Dose Level 2
Started | 3 | 6 | 3 | 3
Completed | 3 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 15 participants with advanced NSCLC
Groups:
- Escalation Arm A Dose Level 1: Patients received trametinib 1.5mg QD and Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm A Dose Level 2: Patients received trametinib 2mg QD and Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm B Dose Level 1: Patients administered Pembrolizumab IV 200 mg IV over 30 minutes. Trametinib dose of 1.5mg QD was given PO on D1-10 starting in course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm B Dose Level 2: Patients administered Pembrolizumab IV 200 mg IV over 30 minutes. Trametinib dose of 2mg QD was given PO on D1-10 starting in course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Escalation Arm A Dose Level 1 | Escalation Arm A Dose Level 2 | Escalation Arm B Dose Level 1 | Escalation Arm B Dose Level 2 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 2 | 0 | 9
  >=65 years | 0 | 2 | 1 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 2 | 9
  Male | 1 | 2 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 2 | 11
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 3 | 2 | 3 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 3 | 3 | 15
Mutation Status [Count of Participants; unit: Participants]
  KRAS G12C | 1 | 0 | 1 | 1 | 3
  KRAS non-G12C | 1 | 6 | 2 | 1 | 10
  BRAF non-V600E | 0 | 0 | 0 | 1 | 1
  RAS Wild Type | 1 | 0 | 0 | 0 | 1
Smoking Status [Count of Participants; unit: Participants]
  Current | 0 | 0 | 0 | 1 | 1
  Former | 3 | 3 | 2 | 2 | 10
  Never | 0 | 3 | 1 | 0 | 4
Prior PD1/PDL1 Treatment [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 2 | 1 | 6
  No | 1 | 5 | 1 | 2 | 9
PD-L1 Expression (TPS 22C3) [Count of Participants; unit: Participants] — Population: PD-L1 expression testing was not done for subject 002 on Arm A, Dose level 1
  Participants
    number analyzed (Participants) | 2 | 6 | 3 | 3 | 14
    0% | 2 | 3 | 3 | 2 | 10
    1-49% | 0 | 3 | 0 | 0 | 3
    >/= 50% | 0 | 0 | 0 | 1 | 1
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 3 | 6 | 3 | 3 | 15
  No | 0 | 0 | 0 | 0 | 0
Prior Immunotherapy [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 2 | 1 | 8
  No | 1 | 3 | 1 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicity (DLT) of Pembrolizumab and Trametinib Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 4.0
Description: The occurrence of toxicities during the first two cycles (i.e. after completion of the lead in cycle and the first cycle where both pembrolizumab and trametinib are administered) will be considered a DLT, if judged by the Investigator to be possibly, probably or definitely related to study drug administration. Adverse events will be summarized descriptively by type and by severity, with number and relative frequency calculated for all non-zero occurrences.
Time Frame: Up to 6 weeks
Population: Overall object is to assess the efficacy of pembrolizumab (MK-3475) when given in combination with trametinib in the proposed sequencing schemes. The data is being reported per Arm as this reflects the difference in the sequencing of Trametinib and Pembrolizumab.
Measure: Number; unit: DLT
Groups:
- Escalation Arm A Dose Level 1: Patients received trametinib 1.5mg QD PO on D1-10. Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm A Dose Level 2: Patients received trametinib 2 mg QD PO on D1-10. Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm B Dose Level 1: Patients administered Pembrolizumab IV 200 mg IV over 30 minutes. Trametinib dose of either 1.5mg QD was given PO on D1-10 starting in course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm B Dose Level 2: Patients administered Pembrolizumab IV 200 mg IV over 30 minutes. Trametinib dose of either 2mg QD was given PO on D1-10 starting in course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Escalation Arm A Dose Level 1 | Escalation Arm A Dose Level 2 | Escalation Arm B Dose Level 1 | Escalation Arm B Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 3
DLT | 0 | 1 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Association with response rate will be summarized descriptively by presenting the mean, standard deviation (SD), and other characteristics of molecular and immune measures, stratified by response status. Will assess whether one arm has superior ORR, using logistic regression analysis to control for clinical covariates.
Time Frame: Up to 3 years
Population: Secondary objective is to evaluate the clinical efficacy of pembrolizumab (MK-3475) when given in combination with trametinib in the proposed sequencing schemes. The data is being reported per Arm as this reflects the difference in the sequencing of Trametinib and Pembrolizumab.
Measure: Number; unit: percentage of participants
Groups:
- Escalation Arm A Dose Level 2: Patients received trametinib 2mg QD PO on D1-10. Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Escalation Arm A Dose Level 1 | Escalation Arm A Dose Level 2 | Escalation Arm B Dose Level 1 | Escalation Arm B Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 3
percentage of participants | 6 | 0 | 0 | 6

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Associations of molecular and immune measures with PFS will be summarized descriptively by stratified Kaplan-Meier curves and, if numbers permit, by proportional hazards models with molecular and immune responses as predictors. Will assess whether one arm has superior PFS, using proportional hazards models to control for clinical covariates.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Escalation Arm A Dose Level 1 | Escalation Arm A Dose Level 2 | Escalation Arm B Dose Level 1 | Escalation Arm B Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 3
months | 4.79 [1.80 to 8.07] | 0 [0 to 0] | 2.08 [1.97 to 2.08] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each patient starting from the first day of study drug administration (D1) and continuing through 30 days after the last dose of the study drug, an average of 5.4 months.
Description: Treatment related adverse events, all grades.
Groups:
- Escalation Arm A Level 1: Patients received trametinib 1.5mg QD PO on D1-10. Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm A Level 2: Patients received trametinib 2mg QD PO on D1-10. Pembrolizumab IV 200 mg IV over 30 minutes was added on day 1 starting with course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm B Level 1: Patients administered Pembrolizumab IV 200 mg IV over 30 minutes. Trametinib dose of 1.5mg QD was given PO on D1-10 starting in course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Escalation Arm B Level 2: Patients administered Pembrolizumab IV 200 mg IV over 30 minutes. Trametinib dose of 2mg QD was given PO on D1-10 starting in course 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Escalation Arm A Level 1 | Escalation Arm A Level 2 | Escalation Arm B Level 1 | Escalation Arm B Level 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 0/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Arm A Level 1 (N=3) | Escalation Arm A Level 2 (N=6) | Escalation Arm B Level 1 (N=3) | Escalation Arm B Level 2 (N=3)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Arm A Level 1 (N=3) | Escalation Arm A Level 2 (N=6) | Escalation Arm B Level 1 (N=3) | Escalation Arm B Level 2 (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (3) | 1 (1) | 1 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
CPK increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03299088/Prot_SAP_000.pdf